CLINICAL TRIAL: NCT01524107
Title: Comparison of Maternal and Fetal Complications After Urgent Caesarian Section for Prolapsed Cord Versus Elective Caesarian Section.
Brief Title: Complications: Urgent C Section VS Elective C Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: CSURGENT-ELECT-HMO-CTIL
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Urgent Caesarian Section Secondary to Cord Prolapse
Keywords: Prophylaxis Antibiotics; Maternal Complications; Neonatal Complications; Cord Prolapse; Elective Caesarian Section; Maternal Morbidity; Neonatal Morbidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urgent Caesarian Section
- Elective Caesarian Section

SUMMARY:
The medical literature does not provide sufficient information or recommendation regarding specific antibiotic coverage for urgent Caesarian sections. The goal of this study is to compare maternal and neonatal morbidity of women who have undergone urgent Caesarian Sections for Prolapsed Cord to those who have undergone Elective Caesarian Sections in order to develop a standard treatment protocol. The Medical Record review will include many parameters including complications, type of antibiotic usage etc.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing urgent Caesarian Section for Prolapsed Cord.
* women undergoing Elective Caesarian Section.

Exclusion Criteria:

* preterm birth
* multiple gestation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing Urgent Caesarian Section for Prolapsed Cord and women undergoing Elective Caesarian Section at Hadassah Medical Center-Har HaTzofim.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner-Celnikier, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel